CLINICAL TRIAL: NCT00793936
Title: Criteria for Choice of Right Double Lumen Tube for Lung Surgery
Brief Title: Criteria for Choice of Right Double Lumen Tube (DLT)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Dr. Gofman Vladislav Senior Anesthesiologist, The Anesthesiology Department, Assaf-Harofeh Medical Center, Israel
Other Study IDs: 160.08
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2008-11-19 (Estimated); Status verified 2008-11

CONDITIONS: Thoracic Surgery
Keywords: Right Double Lumen Tube

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There are specific guidelines for choice of Lt DLT size in correlation to patient's height and tracheal diameter on chest X-ray/CT scan. Accordingly to these criteria the RT DLT size is determined.

Should the criteria for determining the appropriate size be the same for Rt and Lt DLT?

DETAILED DESCRIPTION:
Objective: Adequacy of criteria for Lt DLT size in the determination of RT DLT size before thoracic surgery.

Methods: A prospective, controlled, comparative study. After obtaining informed consent, male and female patients over 18 years of age , candidates for elective thoracic surgery obliging DLT intubation, will be enrolled in the study. Children, pregnant and mentally incompetent patients will not be included.

Preoperative evaluation will be performed by an anesthesiologist and the patients will receive premedication with respect to the planned operation and concurrent disease status. The age, gender, height and weight of the patient will be recorded. On the chest CT series, measurements of the tracheal length and diameter, both main bronchial, and RUL bronchial orifice diameter in millimeters will be performed, using an universal measurement system .

All patients will receive intravenous induction with Fentanyl 3-5 mcg/kg, Propofol 2-2.5 mg/kg, and Rocuronium 0.6-0.8 mg/kg. All patients will be intubated by the same anesthesiologist. Fiberoptic bronchoscopy will be performed for proper positioning of the DLT.

Accordingly to the indication , patients will be intubated with Lt or Rt DLT -Mallinkrodt Broncho-cath, routinely used for this kind of operations.

Patients scheduled for right lung operation will be intubated with Lt DLT. The size of the Lt DLT will be determined accordingly to the guidelines, in correlation with patient's height and CT measurements . Lt DLT intubation will be performed by the generally accepted technique, under FOB control. In case the Lt DLT size will prove to be inappropriate , a smaller/larger DLT will be inserted, accordingly.

Patients scheduled for left lung operation will be intubated with Rt DLT. The size of the Rt DLT will be determined in correlation with patient's height and CT measurements, accordingly to the guidelines for Lt DLT size . In case the Rt DLT positioning is impossible due to inappropriate adjustment of the ventilation slot against the RUL bronchus orifice and/or tracheal protrusion of the bronchial cuff, the Rt DLT will be substituted by a smaller/larger Rt DLT , respectively.

The number of attempts on intubation and repositionings of the DLT during surgery will be recorded.

The volume of air in the bronchial and tracheal cuff will be recorded. Information about the adequacy of lung separation will be obtained by the surgeons.

Postoperative clinical and X-ray follow up will be performed about lung recruitment and ventilatory complications ( atelectasis, pneumonia) Throughout the study no additional x-ray or laboratory checkup will be required, and no additional invasive procedures or treatment will be performed, than the usually accepted.

Statistical analysis of collected clinical and rentgenologic data will be performed .

ELIGIBILITY:
Inclusion Criteria:

* male and female patients over 18 years of age , candidates for elective thoracic surgery obliging DLT intubation, will be enrolled in the study

Exclusion Criteria:

* Children, pregnant and mentally incompetent patients will not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After obtaining informed consent, male and female patients over 18 years of age, candidates for elective thoracic surgery obliging DLT intubation, will be enrolled in the study. Children, pregnant and mentally incompetent patients will not be included.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

REFERENCES:
- [Background] Campos JH, Massa FC, Kernstine KH. The incidence of right upper-lobe collapse when comparing a right-sided double-lumen tube versus a modified left double-lumen tube for left-sided thoracic surgery. Anesth Analg. 2000 Mar;90(3):535-40. doi: 10.1097/00000539-200003000-00007. PMID 10702432
- [Background] Chow MY, Liam BL, Lew TW, Chelliah RY, Ong BC. Predicting the size of a double-lumen endobronchial tube based on tracheal diameter. Anesth Analg. 1998 Jul;87(1):158-60. doi: 10.1097/00000539-199807000-00033. PMID 9661566
- [Background] Benumof JL, Partridge BL, Salvatierra C, Keating J. Margin of safety in positioning modern double-lumen endotracheal tubes. Anesthesiology. 1987 Nov;67(5):729-38. doi: 10.1097/00000542-198711000-00018. PMID 3674473
- [Background] Klein U, Karzai W, Bloos F, Wohlfarth M, Gottschall R, Fritz H, Gugel M, Seifert A. Role of fiberoptic bronchoscopy in conjunction with the use of double-lumen tubes for thoracic anesthesia: a prospective study. Anesthesiology. 1998 Feb;88(2):346-50. doi: 10.1097/00000542-199802000-00012. PMID 9477054
- [Background] Chow MY, Liam BL, Thng CH, Chong BK. Predicting the size of a double-lumen endobronchial tube using computed tomographic scan measurements of the left main bronchus diameter. Anesth Analg. 1999 Feb;88(2):302-5. doi: 10.1097/00000539-199902000-00014. PMID 9972745
- [Background] Amar D, Desiderio DP, Heerdt PM, Kolker AC, Zhang H, Thaler HT. Practice patterns in choice of left double-lumen tube size for thoracic surgery. Anesth Analg. 2008 Feb;106(2):379-83, table of contents. doi: 10.1213/ane.0b013e3181602e41. PMID 18227288
- [Background] Bussieres JS, Lacasse Y, Cote D, Beauvais M, St-Onge S, Lemieux J, Soucy J. Modified right-sided Broncho-Cath double lumen tube improves endobronchial positioning: a randomized study. Can J Anaesth. 2007 Apr;54(4):276-82. doi: 10.1007/BF03022772. PMID 17400979
- [Background] Eberle B, Weiler N, Vogel N, Kauczor HU, Heinrichs W. Computed tomography-based tracheobronchial image reconstruction allows selection of the individually appropriate double-lumen tube size. J Cardiothorac Vasc Anesth. 1999 Oct;13(5):532-7. doi: 10.1016/s1053-0770(99)90003-4. PMID 10527220
- [Background] Hannallah M, Benumof JL, Silverman PM, Kelly LC, Lea D. Evaluation of an approach to choosing a left double-lumen tube size based on chest computed tomographic scan measurement of left mainstem bronchial diameter. J Cardiothorac Vasc Anesth. 1997 Apr;11(2):168-71. doi: 10.1016/s1053-0770(97)90208-1. PMID 9105987
- [Background] Neustein SM. What is the best choice for size of double lumen tube? Anesth Analg. 2008 Jul;107(1):342-3. doi: 10.1213/ane.0b013e318173e773. No abstract available. PMID 18635507